CLINICAL TRIAL: NCT05349097
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study of Orally Administered IMG-004 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Dose(s) and an Open-Label Study of Single Oral Dose of IMG-004 to Evaluate the Food Effect in Healthy Participants
Brief Title: Study to Evaluate IMG-004 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inmagene LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMG-004-101
Record Dates: First submitted 2022-04-17; First posted 2022-04-27 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- SAD cohort 1 active treatment (Experimental): 30mg
  Interventions: Drug: SAD IMG-004 30mg
- SAD cohort 2 active treatment (Experimental): 100mg.
  Interventions: Drug: SAD IMG-004 100mg
- SAD cohort 3 active treatment (Experimental): 200mg
  Interventions: Drug: SAD IMG-004 200mg
- SAD cohort 4 active treatment (Experimental): 400mg.
  Interventions: Drug: SAD IMG-004 400mg
- SAD cohort 5 active treatment (Experimental): 600mg.
  Interventions: Drug: SAD IMG-004 600mg
- SAD cohort 1 placebo (Placebo Comparator): 30mg
  Interventions: Drug: SAD Placebo 30mg
- SAD cohort 2 placebo (Placebo Comparator): 100mg.
  Interventions: Drug: SAD Placebo 100mg
- SAD cohort 3 placebo (Placebo Comparator): 200mg.
  Interventions: Drug: SAD Placebo 200mg
- SAD cohort 4 placebo (Placebo Comparator): 400mg.
  Interventions: Drug: SAD Placebo 400mg
- SAD cohort 5 placebo (Placebo Comparator): 600mg.
  Interventions: Drug: SAD Placebo 600mg
- MAD cohort 1 active treatment (Experimental): 50mg
  Interventions: Drug: MAD IMG-004 50mg
- MAD cohort 1 placebo (Placebo Comparator): 50mg
  Interventions: Drug: MAD Placebo 50mg
- MAD cohort 2 active treatment (Experimental): 150mg
  Interventions: Drug: MAD IMG-004 150mg
- MAD cohort 2 placebo (Placebo Comparator): 150mg
  Interventions: Drug: MAD Placebo 150mg
- MAD cohort 3 active treatment (Experimental): 300mg
  Interventions: Drug: MAD IMG-004 300mg
- MAD cohort 3 placebo (Placebo Comparator): 300mg
  Interventions: Drug: MAD Placebo 300mg
- Food Effect cohort (Experimental): 150mg
  Interventions: Drug: FE IMG-004 150mg

INTERVENTIONS:
Drug: SAD IMG-004 30mg — Each participant will be randomized to receive a single oral dose of 30mg IMG-004
  Arms: SAD cohort 1 active treatment
Drug: SAD IMG-004 100mg — Each participant will be randomized to receive a single oral dose of 100mg IMG-004
  Arms: SAD cohort 2 active treatment
Drug: SAD IMG-004 200mg — Each participant will be randomized to receive a single oral dose of 200mg IMG-004
  Arms: SAD cohort 3 active treatment
Drug: SAD IMG-004 400mg — Each participant will be randomized to receive a single oral dose of 400mg IMG-004
  Arms: SAD cohort 4 active treatment
Drug: SAD IMG-004 600mg — Each participant will be randomized to receive a single oral dose of 600mg IMG-004
  Arms: SAD cohort 5 active treatment
Drug: SAD Placebo 30mg — Each participant will be randomized to receive a single oral dose of 30mg matching placebo
  Arms: SAD cohort 1 placebo
Drug: SAD Placebo 100mg — Each participant will be randomized to receive a single oral dose of 100mg matching placebo
  Arms: SAD cohort 2 placebo
Drug: SAD Placebo 200mg — Each participant will be randomized to receive a single oral dose of 200mg matching placebo
  Arms: SAD cohort 3 placebo
Drug: SAD Placebo 400mg — Each participant will be randomized to receive a single oral dose of 400mg matching placebo
  Arms: SAD cohort 4 placebo
Drug: SAD Placebo 600mg — Each participant will be randomized to receive a single oral dose of 600mg matching placebo
  Arms: SAD cohort 5 placebo
Drug: MAD IMG-004 50mg — Each participant will be randomized to receive daily oral dose of 50mg IMG-004 for 10 days
  Arms: MAD cohort 1 active treatment
Drug: MAD Placebo 50mg — Each participant will be randomized to receive daily oral dose of 50mg matching placebo for 10 days
  Arms: MAD cohort 1 placebo
Drug: MAD IMG-004 150mg — Each participant will be randomized to receive daily oral dose of 150mg IMG-004 for 10 days
  Arms: MAD cohort 2 active treatment
Drug: MAD Placebo 150mg — Each participant will be randomized to receive daily oral dose of 150mg matching placebo for 10 days
  Arms: MAD cohort 2 placebo
Drug: MAD IMG-004 300mg — Each participant will be randomized to receive daily oral dose of 300mg IMG-004 for 10 days
  Arms: MAD cohort 3 active treatment
Drug: MAD Placebo 300mg — Each participant will be randomized to receive daily oral dose of 300mg matching placebo for 10 days
  Arms: MAD cohort 3 placebo
Drug: FE IMG-004 150mg — A single dose of IMG-004 at 150 mg dose level will be administered to the participants in fed and fasted states
  Arms: Food Effect cohort

SUMMARY:
A Phase 1, Randomized, Double-blind, Placebo-controlled Study of Orally Administered IMG-004 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Dose(s) and an Open-Label Study of Single Oral Dose of IMG-004 to Evaluate the Food Effect in Healthy Participants

DETAILED DESCRIPTION:
The study is a Phase 1, randomized, double-blind, placebo-controlled study of orally administered IMG-004 to evaluate the safety, tolerability, and pharmacokinetics of single and multiple ascending doses in healthy participants, in which 8 dosing cohort levels are planned to be evaluated. Food Effect of IMG-004 will also be evaluated in single oral dose of IMG-004 in healthy participants

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females, 18 to 60 years of age (inclusive) at the date of signed consent form.
2. Body mass index (BMI) greater than or equal to 18.5 and less than 32 (kg/m2) and a minimum body weight of 45 kg.
3. Able to participate and comply with all study procedures and restrictions, and willing to provide written informed consent to participate in the study.
4. Male participants must agree to practice true abstinence; be surgically sterilized (performed at least 6 months prior and documented to no longer produce sperm - verbal confirmation through medical history review acceptable); or agree to use a condom plus ensure use of effective contraception by their female partner of childbearing potential (ie, established use of hormonal contraception - started at least 30 days before Day 1; or placement or an intrauterine device or intrauterine system, diaphragm with spermicide or cervical sponge with spermicide) from screening and for at least 30 days after dosing and refrain from donating sperm during this period. Contraception requirements do not apply for participants in an exclusively same-sex relationship or if their female partner is of non-childbearing potential. Males with pregnant partners may participate if they agree to use a barrier method of contraception.
5. Female participants of non-childbearing potential, defined as surgically sterile (hysterectomy, bilateral salpingectomy, bilateral tubal ligation or bilateral oophorectomy, verbal confirmation through medical Confidential Page 17 of 75 history review acceptable) or postmenopausal (no menses for 12 months and confirmed by follicle-stimulating hormone (FSH) level ≥ 40 mIU/mL).

Exclusion Criteria:

1. History of disease of the central nervous system, cardiovascular system, kidney, liver, digestive system, respiratory system, or metabolic/endocrine system, or other disease that in the opinion of the Investigator (or medically qualified designee) may make participation unsafe for the participant or interfere with trial evaluations or otherwise considered clinically significant.
2. History of immunological abnormality (eg, primary or secondary immune suppression) that in the opinion of the Investigator (or medically qualified designee) may make participation unsafe for the participant or interfere with trial evaluations or otherwise considered clinically significant.
3. History of severe immediate hypersensitivity reaction to BTK inhibitors, defined as non-cutaneous hypersensitivity reaction, requiring parenteral (IM/IV) therapy.
4. Major surgery ≤ 4 weeks before Baseline visit. Participants must have also fully recovered from any surgery (major or minor) and/or its complications before initiating study treatment.
5. History of malignancy or known current malignancy, except for adequately treated basal cell or squamous cell carcinoma of the skin.
6. Participants who, in the Investigator's judgement, are perceived as having an increased risk of bleeding, eg, history of hemorrhagic disorders, clinical relevant petechial bleeding, occult blood in feces, hematuria in repeated urine tests(unless attributed to menstruation), trauma or surgery within the last month, planned surgery during trial participation, history of arteriovenous malformation or aneurysm, history of gastroduodenal ulcer disease or gastrointestinal hemorrhage, history of intracranial, intraocular, spinal, retroperitoneal, or atraumatic intraarticular bleeding, use of drugs that may interfere with hemostasis during trial conduct (eg, acetylic salicylic acid or other non-steroidal anti-inflammatory drugs)
7. Participant has an active infection or history of infections as follows:

   1. Acute infection requiring treatment with oral antibiotics, anti-virals, anti-parasitics, anti-protozoal, or anti-fungals within 14 days before the Baseline visit.
   2. A serious infection, defined as requiring hospitalization or intravenous anti-microbial therapy within 2 months prior to Baseline visit.
   3. A history of opportunistic, recurrent, or chronic infections.
8. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or antibody to Hepatitis B core antigen (HBcAb) with positive test for HBV DNA (> 500 IU/ml) or hepatitis C antibodies (HCV) at Screening visit.
9. Having evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB) as defined by the following:

   1. Positive Interferon Gamma Release Assay (IGRA) (with one of the following acceptable assays: QuantiFERON(R)-TB Gold (QFT-G) test, T-SPOT TB, QuantiFERON-TB Gold In-Tube test (QFT-GIT)) performed during Screening or within 3 months prior to Day 1. OR
   2. History of either untreated or inadequately treated latent or active TB infection.
10. Participants with positive testing for COVID-19 at the Baseline visit.
11. Participants with clinically significantly abnormal laboratory values, as determined by the Investigator (or medically qualified designee), including but not limited to:

    1. Absolute neutrophil count ≤ 1,500/μL or absolute lymphocyte count ≤ 800/μL, or eosinophil count > 700/μL, platelet counts < 100 × 109/L, hemoglobin < ULN, or any abnormal evaluations judged clinically significant by the Investigator (or medically qualified designee) at the Screening or Baseline visits. A single repeat of laboratory tests is permissible at Screening and Baseline, if deemed required by PI or medically qualified designee.
    2. Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≥ values of more than 1.5 times the upper limit of normal (ULN), which remains similar upon repeat, at the Screening or Baseline visits.
    3. Total bilirubin above ULN, which remains similar upon repeat, at the Screening or Baseline visits.
    4. Participants with Creatinine clearance rate < 80 mL/min as determined by the Cockcroft Gault formula, which remains similar upon repeat, at the Screening or Baseline visits.
12. Closure time testing or platelet aggregometry testing (to monitor platelet function) outside of reference range at Screening or Baseline visit.
13. QTcF greater than 450 msec (males) or greater than 470 msec (females) at Screening or Baseline visit (if out of range, repeat twice and average the 3 readings for eligibility purposes) or deemed clinically significant by the Investigator (or medically qualified designee).
14. Screening ECG with QRS and/or T-wave judged to be unfavorable for a consistently accurate QT measurement as judged by the Investigator (or medically qualified designee).
15. Clinically significant abnormal screening values in clinical (electrocardiograms [ECGs], vital signs, physical examination) and laboratory tests in the opinion of the Investigator (or medically qualified designee). Up to two repeats of assessments or tests can be conducted at the discretion of the Investigator (or medically qualified designee).
16. Use of any prescription medication within the 14 days prior to the first study drug administration or five half-lives, whichever is longer.
17. Use of over-the-counter medication within 7 days prior to the first study drug administration, including herbal medicines, that in the opinion of the Investigator (or medically qualified designee) may make participation unsafe for the participant or interfere with trial evaluations.
18. Average alcohol consumption of more than 14 units/week for females and 21 units/week for males (1 unit = one half-pint beer, 25 mL of 40% spirit or a 125-mL glass of wine).
19. Use of more than 5 tobacco/nicotine-containing products per month within 6 months prior to the IMP administration.
20. History of, or current substance abuse considered significant by the Investigator (or medically qualified designee) or positive urine drug and alcohol breath (or urine alcohol) testing at the Screening or Baseline visits.
21. Live (attenuated) vaccination within 8 weeks before Screening visit or plan to be vaccinated by live (attenuated) vaccine during the trial (until completion of the final follow-up visit).
22. COVID-19 vaccination, or influenza vaccination (inactivated), within 14 days prior to IMP administration or planning to receive COVID-19 vaccination or influenza vaccination (inactivated) within 14 days post IMP administration.
23. Receipt of an investigational drug or medical device within 30 days or 5 half-lives (whichever is longer) prior to Day 1 dosing.
24. Donated or lost more than 500 mL of blood or plasma within 3 months of the Screening visit or received blood products within 8 weeks of the Screening visit.
25. Participant has a disease that might affect drug absorption, distribution, metabolism, and excretion based on the Investigator (or medically qualified designee)'s judgement (eg, gastrointestinal dysfunction, peptic ulcer, gastrointestinal surgery [except appendectomy and uncomplicated hernia repair], etc.)
26. Cannot communicate adequately in English or cannot commit to full participation in all trial procedures.
27. Pregnant or lactating women.
28. Inability to comply with dietary regimen of the trial site.
29. Any other circumstances that, in the Investigator (or medically qualified designee)'s judgment, may increase the risk associated with the participant's participation in and completion of the study or could preclude the evaluation of the participant's response.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Safety of IMG-004 | SAD cohort from signing ICF up to Day 15; MAD cohort: from signing ICF to Day24
  Incidence and severity of AEs, including clinically relevant findings from vital signs, physical examination, laboratory tests, and 12-lead ECG

SECONDARY OUTCOMES:
PK parameters of IMG-004 | SAD cohort from day 1 to day 8, MAD cohort from day 1 to day 17, FE cohort from day 1 to day 8
  Single Dose: Cmax, Tmax, AUClast, etc. Multiple dose: Cmax-ss), Tmax-ss, AUCss, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Cru, Daytona Beach, Florida, United States